CLINICAL TRIAL: NCT01102452
Title: A Randomized, Two-Regimen, Crossover, Comparative Study to Evaluate the Blood Glucose Regulation and Safety of PPB-R-203-02 Based Noodle Versus Commercially Available Wet Noodle in 24 Patients With Diabetes
Brief Title: A Study to Evaluate the Blood Glucose Regulation and Safety of PPB-R-203-02 Based Noodle Versus Commercially Available Wet Noodle in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharma Power Biotec Co., Ltd. (Industry)
Responsible Party: isRed Pharma & Biotech Research Corporation, Isredbioresearch
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: PPB-R-203-02
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2010-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Commercially Available Wet Noodle (Placebo Comparator): Commercially Available Wet Noodle will be served as a diet equivalent to daily energy needs as judged by indirect calorimetry and of same macronutrient composition.
  Interventions: Dietary Supplement: Commercially Available Wet Noodle
- PPB-R-203-02 Noodle (Experimental): PPB-R-203-02 Noodle is manufacture by Pharma Power Biotec Co., Ltd. The composition of PPB-R-203-02 Noodle is resistant starch (RS). By definition, resistant starch (RS) is any starch that is not digested in the small intestine but passes to the large intestine (or the colon). Therefore, resistant starch can be regarded as a component of dietary fiber. PPB-R-203-02 Noodle will be served as a diet equivalent to daily energy needs as judged by indirect calorimetry and of the same macronutrient composition.
  Interventions: Dietary Supplement: PPB-R-203-02 Noodle

INTERVENTIONS:
Dietary Supplement: Commercially Available Wet Noodle — Commercially Available Wet Noodle will be served as a diet equivalent to daily energy needs as judged by indirect calorimetry and of same macronutrient composition.
  Arms: Commercially Available Wet Noodle
Dietary Supplement: PPB-R-203-02 Noodle — PPB-R-203-02 Noodle is manufacture by Pharma Power Biotec Co., Ltd. The composition of PPB-R-203-02 Noodle is resistant starch (RS). By definition, resistant starch (RS) is any starch that is not digested in the small intestine but passes to the large intestine (or the colon). Therefore, resistant starch can be regarded as a component of dietary fiber. PPB-R-203-02 Noodle will be served as a diet equivalent to daily energy needs as judged by indirect calorimetry and of the same macronutrient composition.
  Arms: PPB-R-203-02 Noodle

SUMMARY:
To evaluate the result of PPB-R-203-02 based noodle and commercially available wet noodle on blood glucose control in 24 patients with diabetes for 2 days.

DETAILED DESCRIPTION:
The MiniMed Medtronic CGMS (continuous glucose monitoring system), the first model approved by FDA, was used for subcutaneous glucose monitoring. The CGMS continually measures the glucose concentration of the interstitial fluid every 10 seconds and then stores an average glucose value for each 5 minutes period, for a total of up to 288 measurements each day.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus patient.
2. Aged between 20 to 65 years old.
3. Informed consent form signed.

Exclusion Criteria:

1. A recent history of drug or alcohol abuse.
2. Sensitivity to analogous product.
3. Serious cardiovascular disorders.
4. Participation in another clinical investigation study.
5. Ongoing influenza, autoimmune disease and other metabolic diseases.
6. Pregnant or lactating women.
7. Individuals are judged by the investigators or co-investigator to be undesirable as subjects.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The daily blood glucose level will be monitored by the CGMS (continuous glucose monitoring system)device | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- PingTung Christian Hospital, Pingtung City, Taiwan